CLINICAL TRIAL: NCT07203417
Title: A Randomized Trial Comparing a Sex Education and Therapy Online Intervention Delivered With and Without Professional Guidance for the Treatment of Sexual Desire Discrepancy in Couples
Brief Title: Evaluating Sexual Psychoeducation in Couples With Sexual Desire Discrepancy
Acronym: STEP for SDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lori Brotto, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MFE-193938
Record Dates: First submitted 2025-09-20; First posted 2025-10-02 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-09

CONDITIONS: Sexual Desire
Keywords: Psychoeducation; Sex Therapy; Online Intervention; Dyadic Treatment
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: This is a parallel-assignment interventional study with three arms: STEP-T, STEP-NT, and Waitlist. Participants are initially randomized to one of these three arms. After 10 weeks, participants in the Waitlist arm are re-randomized to either STEP-T or STEP-NT. STEP-T and STEP-NT participants continue their assigned interventions without crossover. This design allows us to determine that improvements in clinical outcomes are due to the STEP intervention rather than the mere passage of time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STEP-T (Active Comparator): Participants assigned to this arm will receive STEP guided by a therapist.
  Interventions: Behavioral: STEP-T
- STEP-NT (Active Comparator): Participants assigned to this arm will receive STEP without therapist guidance.
  Interventions: Behavioral: STEP-NT
- Waitlist (Other): Participants in this arm will not receive any treatment during the first 10 weeks. After 10 weeks, the participants in this arm are re-randomized to either STEP-T or STEP-NT.
  Interventions: Other: Waitlist

INTERVENTIONS:
Behavioral: STEP-T — Couples in the STEP-T group will meet online with a therapist for 120 minutes once a week over 8 weeks. Each meeting consists of a therapist-led session focused on the psychoeducational content from the STEP module. Sessions begin with a review of the homework completed during the previous week and end with the assignment of new sex therapy homework related to that day's session. After each session, the therapist will email the couple the module that includes the session's psychoeducational handouts and the sex therapy homework to be completed prior to the next session.
  Arms: STEP-T
Behavioral: STEP-NT — Couples in the STEP-NT group will receive STEP (i.e., one module per week for 8 weeks, including psychoeducational handouts and sex therapy homework), without the therapist-led online sessions. However, like couples in STEP-T, they will be allowed to contact the research team for clarifications related to the structure, instructions, or technical aspects of the exercises. This support will be limited to non-clinical guidance and will not involve any individualized feedback regarding participants' personal experiences or relationship dynamics.
  Arms: STEP-NT
Other: Waitlist — While couples randomized to STEP-T and STEP-NT will complete one online baseline assessment battery before randomization, those assigned to the waitlist control condition will complete two baseline assessments online, spaced 10 weeks apart, before being randomized to one of the active treatment groups (i.e., STEP-T or STEP-NT). The 10-week waiting period was selected to match the time it takes couples to complete the 8 modules of STEP. This design allows us to determine that improvements in clinical outcomes are due to the STEP intervention rather than the mere passage of time. Following the post-waiting period assessment (i.e., the second baseline battery), waitlist participants will be randomized to STEP-T or STEP-NT.
  Arms: Waitlist

SUMMARY:
Sexual desire discrepancy (SDD) occurs when partners have different levels of sexual desire and are distressed by it. It is one of the most common reasons couples seek help, but no proven dyadic treatment currently exists. This study will test STEP, an online program designed to support couples with SDD. The investigators will compare two formats of STEP: one with therapist support and one self-guided, against a waitlist control group. The investigators will also assess how satisfied couples are and how they engage with the two online formats. This study will generate new data on how effective STEP is with and without guidance, and inform treatment guidelines.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of an 8-week online intervention (STEP) designed to reduce distress related to SDD in couples. Two formats of the intervention will be tested: a therapist-guided version (STEP-T) and a self-guided version (STEP-NT). Couples will be randomly assigned to one of these formats or to a waitlist control group.

The study will assess whether both versions of STEP reduce SDD and associated distress, and whether improvements are maintained over a 6-month follow-up. The investigators will also examine participants' satisfaction with the program, engagement, and retention rates.

In addition, the investigators will explore the psychological factors (e.g., quality of sexual communication, emotional intimacy, interoceptive awareness, and self-compassion) that may explain how the intervention works, as well as whether its effectiveness varies based on relationship duration and participants' perceptions of the treatment's credibility.

Finally, the study will gather exploratory information about potential contributing factors to SDD and how couples experience desire-related challenges, using structured worksheets.

The investigators hypothesize that: a) Both STEP-T (therapist-guided) and STEP-NT (self-guided) will significantly reduce sexual desire discrepancy (SDD) and related distress, compared to a waitlist control group; b) Participants in both intervention groups will show improvements in sexual satisfaction, relationship satisfaction, and sexual pleasure; c) These improvements will be maintained at 6-month follow-up; d) STEP-T will produce greater improvements than STEP-NT; e) Participants will report moderate to high satisfaction, consistent homework engagement, and retention rates above 70%, with higher engagement expected in the STEP-T group; f) Increases in interoceptive awareness, emotional intimacy, and sexual communication will predict improvements in SDD and distress. Improvements in self-compassion will predict reduced distress; g) Longer relationship duration and higher perceived treatment credibility will be associated with better outcomes.

Once both members of the couple have consented to participate in the study, they will be emailed a Qualtrics link to individually complete a baseline battery of questionnaires (Time 1) and their alphanumerical code to both keep their answers confidential and make researchers able to associate their answers for statistical purposes. In the baseline battery of questionnaires, participants will complete demographic questions (e.g., age, marital status), measures assessing primary and secondary outcomes, measures of mediators, and of relationship duration (moderator). Once completed, participants will be randomized to STEP-T, STEP-NT, or a waitlist control condition. Participants will be informed about which treatment type they were randomized to via e-mail. Couples initially randomized to the waitlist will complete a second baseline battery of questionnaires (including the same measures of the first baseline battery) after a 10-week waiting period. No treatment will be given to waitlist participants during this waiting period. After this period, they will be randomized to either STEP-T or STEP-NT and will be informed about which treatment type they were randomized to via e-mail.

After scheduling the start date of the treatment, couples in the STEP-T group will meet online with the therapist via videoconferencing software (secure university Zoom account) for 120 minutes/week for 8 weeks. Couples in the STEP-NT group will also have their treatment start date scheduled and will receive one self-guided module per week via email over the course of 8 weeks. Treatment for both groups will begin within one week following the completion of the baseline assessment battery. Participants in both STEP-T and STEP-NT will individually complete, immediately before the start of the next module (for STEP-NT)/session(for STEP-T), an online measure and a homework checklist assessing their engagement with the previously completed module.

In the event that a session (STEP-T) or a module (STEP-NT) is rescheduled, it will preferably be made up within the same week it was originally planned. If that is not possible, the session/module will be made up the following week, in order to minimize the impact on the overall program schedule. Couples in STEP-T will complete treatment credibility measure immediately after session 1 while those in STEP-NT will complete it immediately before receiving module 2. Before Session 3, both members of the couple will be asked to email their completed 3P and Basson's sexual response model worksheets. Before Session 4, both members of the couple will be asked to email their sexual beliefs worksheets. Before Session 5, participants will be asked to email their CBT diamond worksheets and their biases worksheets. Time 1 and an additional questionnaire (measure of treatment satisfaction) will be readministered 2-4 weeks after treatment (Time 2), and again at 6-month follow-up (Time 3; except measure of treatment satisfaction).

The study will be administered entirely online. The research team will follow up with participants who do not respond to emails, fail to complete questionnaires, or miss a session without prior notice, sending up to three reminder emails. If participants do not respond after three follow-up attempts, they will be excluded from the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be a couple;
2. Be in a romantic relationship for at least one year;
3. Be 19 years of age or older;
4. Experience perceived and/or actual SDD with personal and/or relational distress reported by at least one partner;
5. Be fluent in English;
6. Be willing to participate in 8 weekly online treatment sessions;
7. For couples in long-distance relationships, be able to meet the partner in person and via video call to complete the couple's homework;
8. Be willing to abstain from starting any new treatment for SDD for the duration of the study;
9. Be willing to voluntarily complete questionnaires administered before, during, and after the treatment;
10. Have access to an electronic device capable of running Zoom platform (if randomized to STEP-T);
11. Have a stable internet connection.

Exclusion Criteria:

1. Cases where the discrepancy is attributable to at least one partner identifying as asexual (asexuality is not considered a sexual dysfunction; APA, 2013);
2. Presence of untreated psychiatric conditions at the time of recruitment (e.g., depression) that would interfere with participating in the treatment and homework;
3. Receive dyadic psychosexual treatment for SDD elsewhere during the study period.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
A change in relational sexual distress | At baseline (T1), post-treatment (2-4 weeks after STEP completion; T2), and 6-month follow-up (T3).
  Relational sexual distress will be measured using the 6-item Relational Concern subscale of the 30-item Sexual Satisfaction Scale (SSS; Meston & Trapnell, 2005).
A change in personal sexual distress | At baseline (T1), post-treatment (2-4 weeks after STEP completion; T2), and 6-month follow-up (T3).
  Personal sexual distress will be measured using the 13-item Female Sexual Distress Scale-Revised (female version: FSDS-R; Derogatis et al., 2008; male version: Santos-Iglesias et al., 2018).
A change in perceived sexual desire discrepancy | At baseline (T1), post-treatment (2-4 weeks after STEP completion; T2), and 6-month follow-up (T3).
  Perceived sexual desire discrepancy will be measured by asking participants questions on their personal desire and their personal perception of partner's desire. Personal desire will be assessed by the 7-item Partner-related sexual desire subscale of the 13-item SDI-2 (Castro-Calvo et al., 2024). The personal perception of partner's desire will be measured by adapting the original version of SDI-2. SDD will be calculated by doing the absolute difference between one's personal desire and the personal perception of partner's desire scores.
A change in actual sexual desire discrepancy | At baseline (T1), post-treatment (2-4 weeks after STEP completion; T2), and 6-month follow-up (T3).
  The actual sexual desire discrepancy will be measured by calculating the absolute difference between both partners' personal desire scores. Personal desire will be assessed by the 7-item Partner-related sexual desire subscale of the 13-item SDI-2 (Castro-Calvo et al., 2024).

SECONDARY OUTCOMES:
A change in sexual satisfaction | At baseline (T1), post-treatment (2-4 weeks after STEP completion, T2), and 6-month follow-up (T3).
  Sexual satisfaction will be measured by the 20-item The New Sexual Satisfaction Scale (NSSS; Stulhofer et al., 2010).
A change in relational satisfaction | At baseline (T1), post-treatment (2-4 weeks after STEP completion, T2), and 6-month follow-up (T3).
  Relational satisfaction will be measured using the 7-item Relationship Satisfaction Scale (RAS; Hendrick et al., 1998).
A change in sexual pleasure | At baseline (T1), post-treatment (2-4 weeks after STEP completion, T2), and 6-month follow-up (T3).
  Sexual pleasure will be measured using the Experiences of Sexual Pleasure Scale (ESPS; Jabs & Brotto, manuscript in preparation).
Treatment satisfaction | At post-treatment (2-4 weeks after STEP completion, T2).
  Treatment satisfaction will be measured by the 11-item Erectile Dysfunction Inventory of Treatment Satisfaction - Patient Version (Patient EDITS; Althof et al., 1999; adapted for use with a dyadic sample with SDD).

OTHER OUTCOMES:
Mediator through which STEP-T and STEP-NT improve the primary endpoints (self-compassion/self-criticism) | At baseline (T1), post-treatment (2-4 weeks after STEP completion, T2), and 6-month follow-up (T3).
  Self-compassion/self-criticism will be measured by the 26-item Self-Compassion Scale (Costa et al., 2016).
Mediator through which STEP-T and STEP-NT improve the primary endpoints (Interoceptive awareness) | At baseline (T1), post-treatment (2-4 weeks after STEP completion, T2), and 6-month follow-up (T3).
  Interoceptive awareness will be measured by the 37-item Multidimensional Assessment of Interoceptive Awareness (MAIA-2; Mehling et al., 2018).
Mediator through which STEP-T and STEP-NT improve the primary endpoints (Emotional Intimacy) | At baseline (T1), post-treatment (2-4 weeks after STEP completion, T2), and 6-month follow-up (T3).
  Emotional Intimacy will be assessed using the 6-item Emotional Intimacy subscale of the Personal Assessment of Intimacy in Relationships Inventory (PAIR Inventory; Schaefer & Olson, 1981).
Mediator through which STEP-T and STEP-NT improve the primary endpoints (Quality of sexual communication) | At baseline (T1), post-treatment (2-4 weeks after STEP completion, T2), and 6-month follow-up (T3).
  Quality of sexual communication will be assessed using the 13-item Dyadic Sexual Communication Scale (DSCS; Catania, 2013).
Moderator of the treatment effects (relationship duration) | At baseline (T1).
  Relationship duration will be assessed by one ad-hoc question asking participants to report relationship duration in years ("Please indicate the length of your current relationship in years").
Moderator of the treatment effects (treatment credibility) | In STEP-T: Immediately after Session 1. In STEP-NT: Before receiving module 2.
  Treatment credibility will be evaluated with two items as in Brotto et al., 2021; 2022: "To what extent do you think the treatment you will receive is logical in terms of alleviating your couple's sexual desire discrepancy?" and "To what extent do you expect improvement in your couple's sexual desire discrepancy as a result of this treatment?".
Homework engagement | HRS and Homework Checklist: Immediately before each next session/module. Global Homework Checklist: At post-treatment (2-4 weeks after STEP completion, T2) and 6-month follow-up (T3).
  Homework engagement will be measured by the Homework Rating Scale (HRS; Kazantzis et al., 2005), the Homework Checklist, and the Global Homework Checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Brotto, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - UBC Sexual Health Lab, Vancouver Hospital, Vancouver, British Columbia
  - University of British Columbia, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) for this study, due to the sensitive nature of couple-level data and the associated risk of re-identification.

REFERENCES:
- [Background] Marieke D, Joana C, Giovanni C, Erika L, Patricia P, Yacov R, Aleksandar S. Sexual Desire Discrepancy: A Position Statement of the European Society for Sexual Medicine. Sex Med. 2020 Jun;8(2):121-131. doi: 10.1016/j.esxm.2020.02.008. Epub 2020 Mar 16. PMID 32192965
- [Background] Brotto LA, Zdaniuk B, Chivers ML, Jabs F, Grabovac AD, Lalumiere ML. Mindfulness and Sex Education for Sexual Interest/Arousal Disorder: Mediators and Moderators of Treatment Outcome. J Sex Res. 2023 May;60(4):508-521. doi: 10.1080/00224499.2022.2126815. Epub 2022 Sep 30. PMID 36178481
- [Background] Brotto LA, Zdaniuk B, Chivers ML, Jabs F, Grabovac A, Lalumiere ML, Weinberg J, Schonert-Reichl KA, Basson R. A randomized trial comparing group mindfulness-based cognitive therapy with group supportive sex education and therapy for the treatment of female sexual interest/arousal disorder. J Consult Clin Psychol. 2021 Jul;89(7):626-639. doi: 10.1037/ccp0000661. PMID 34383535